CLINICAL TRIAL: NCT00923572
Title: Yasmin Regulatory Post Marketing Surveillance
Brief Title: Yasmin Post Marketing Surveillance
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 14339; YA0510KR (Other: company internal)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Contraception
Keywords: Oral contraceptive
MeSH Terms: interventions — drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: EE30/DRSP (Yasmin, BAY86-5131)

INTERVENTIONS:
Drug: EE30/DRSP (Yasmin, BAY86-5131) — Patients in daily life clinical practice treatment receiving Yasmin according to indication on the label.

SUMMARY:
The objective of this Post Marketing Surveillance (PMS) is to gain information about safety and efficacy in real practice.

ELIGIBILITY:
Inclusion Criteria:

* Women who need oral contraceptive

Exclusion Criteria:

* Patient who belongs to contraindication listed on the product label.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Korean women who need oral contraceptive
Sampling Method: Non-Probability Sample
Enrollment: 777 (Actual)
Dates: Start 2007-12; Primary Completion 2013-05 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Safety and efficacy in real practice | After 6 cycle of treatment

SECONDARY OUTCOMES:
Demography | At initial visit
Medical History | At initial visit
Administration period of Yasmin | After 6 cycle of treatment or at the point of withdrawan
Patient's compliance | After 6 cycle of treatment or at the point of withdrawan
Adverse Event / Serious AE collection | At point of the occurence

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, South Korea